CLINICAL TRIAL: NCT06680947
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIb, Effcacy and Safety Study of Recombinant Anti-IL-5 Humanized Monoclonal Antibody Therapy in Adult Subjects With Severe Asthma
Brief Title: A Phase IIb Study of 610 in Participants With Severe Eosinophilic Asthma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-610-BA-II-02
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Subjects will receive 610 for 52 weeks.
  Interventions: Drug: 610
- Group B (Experimental): Subjects will receive 610 for 52 weeks.
  Interventions: Drug: 610
- Placebo group (Placebo Comparator): Subjects will receive placebo for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 610 — Subcutaneously injection.
  Arms: Group A
Drug: 610 — Subcutaneously injection.
  Arms: Group B
Drug: Placebo — Subcutaneously injection.
  Arms: Placebo group

SUMMARY:
This study will assess the effcacy and safety of 610 as an adjunctive therapy in adult subjects with severe eosinophilic asthma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the effcacy and safety of 610 in adults with severe eosinophilic asthma. Subjects divided into 3 groups: A group,B group and placebo group. The study is divided into screening period of 4 weeks, treatment period of 16 weeks, prolonged treatment period of 36 weeks and follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and follow the protocol requirements, and give written informed consent prior to participation voluntarily in the study.
* 2. Female and male aged 18 to 75 years.
* 3. Diagnosed with asthma for ≥12 months that meet GINA.
* 4. History of physician-diagnosed asthma requiring treatment with ICS and at least one other control medication for at least 6 months prior to screening.
* 5. Documented history of ≥ 1 moderate exacerbations within 12 months prior to screening.
* 6. Asthma Control Questionnaire question version (ACQ) score ≥1.5 at the screening visit and the randomization visit.

Exclusion Criteria:

* 1. Presence of a known pre-existing, clinically important lung condition other than Asthma.
* 2. Severe asthma exacerbation within 4 weeks prior to randomization.
* 3. Subjects with any eosinophilic diseases other than asthma.
* 4. Known, pre-existing severe or clinically significant cardiovascular disease.
* 5. known, pre-existing other concurrent clinically significant medical conditions that are uncontrolled with standard treatment.
* 6. Subjects who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
* 7. Subjects with allergy/intolerance to a monoclonal antibody.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) at week 52 | Baseline (Day 1) and at week 52
  FEV1 is defined as the volume of air expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry.

SECONDARY OUTCOMES:
Changes from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) at week 16 | Baseline (Day 1) and at week 16
  FEV1 is defined as the volume of air expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry.
Percentage change from baseline in pre-bronchodilator FEV1 at weeks 4, 8,12,16, 20, 28, 36, 44, 52 | Baseline (Day 1) and at week 4, 8,12,16, 20, 28, 36, 44, 52
  Percentage of FEV1 will be measured using spirometry.
Number of asthma exacerbation through study week 52 | From baseline (Day 1) to week 52
  Annualized rate of severe exacerbation events during the 52-week placebo-controlled treatment period
Number of asthma exacerbations requiring hospitalization or emergency room visits | From baseline (Day 1) to week 52
  Asthma exacerbations that are associated with a hospitalization or an emergency room visit.
Change from baseline in Asthma Control Questionnaire (ACQ) score. | From baseline (Day 1) to week 52
  The ACQ contains five symptom questions (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze), one bronchodilator question and pre-bronchodilator FEV1 level. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ score is the average of the responses. Higher score indicates more limitations.
Change from baseline in ST. GEORGE'S Respiratory Questionnaire(SGRQ) | From baseline (Day 1) to week 52
  The SGRQ is designed to measure health impairment in patients with asthma and COPD. It contains two parts: Part 1 (Questions 1 to 8) covers the patients' recollection of their symptoms over a preceding 4 weeks; Part 2, 42 items, relates to the daily activity and psychosocial impacts of the individual's respiratory condition. Total score is presented as a percentage of overall impairment, in which 100 represents the worst possible health status, while 0 indicates the best.
Assessment of adverse events (AEs) | Up to week 60
  Number of participants with adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhang, Doctor, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China